CLINICAL TRIAL: NCT06306430
Title: Detection of Lipoarabinomannan in Urine, Evaluation of the STANDARDTM F TB LAM FIA and Its Impact on the Initial Diagnosis of TB
Brief Title: Detection of Lipoarabinomannan in Urine Evaluation of the STANDARDTMF TBLAMFIA and Its Impact on the Initial TB Diagnosis
Acronym: uLAMTBFIA
Status: Not yet recruiting | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Daniela Maria Cirillo, head Emerging Bacterial Pathogens Unit, Ospedale San Raffaele
Other Study IDs: uLAM TB FIA
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-05

CONDITIONS: Tuberculosis; Diagnoses Disease
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PTB: Subjects with a pulmonary TB
  Interventions: Device: STANDARDTM F TB LAM FIA
- PNTM: Subjects with pulmonary NTM
  Interventions: Device: STANDARDTM F TB LAM FIA
- extraPTB: Subjects with extrapulmonary TB
  Interventions: Device: STANDARDTM F TB LAM FIA
- HC: Healthy controls donors
  Interventions: Device: STANDARDTM F TB LAM FIA

INTERVENTIONS:
Device: STANDARDTM F TB LAM FIA — STANDARDTM F TB LAM Ag FIA is a fluorescent immunoassay for the qualitative detection of specific antigen from mycobacterial lipoarabinomannan (LAM) in urine specimen. STANDARDTM F TB LAM Ag FIA should be used with the STANDARD F Analyzers manufactured by SD BIOSENSOR.

SUMMARY:
Evaluation of the performance of an in vitro test, the STANDARDTM F TB LAM Ag FIA (SD BIOSENSOR, INC.) for the early diagnosis of tuberculosis (TB) infection. This test is for in vitro professional diagnostic use and intended as an aid to early diagnosis of tuberculosis infection. The test will be used according to the instructions for use (IFU).

DETAILED DESCRIPTION:
STANDARDTM F TB LAM Ag FIA is a fluorescent immunoassay which detects lipoarabinomannan in human urine sample. The test evaluated in this study may provide benefits for the development of non sputum-based, less invasive tuberculosis diagnostics that include easier to collect biological samples. The study can therefore be relevant for updating WHO guidelines for TB diagnosis. The results of the STANDARDTM F TB LAM Ag FIA will be interpreted according to the manufacturer´s instructions and will be compared to the results of the test performed to confirm the pulmonary TB, the extrapulmonary TB or the pulmonary NTM diagnosis (intention to treat assay). The test will be repeted at the end of the anti-TB therapy to evaluate if the test can be used as marker of treatment response. Healthy subjects without exposure or risk for TB factors will serve as a proxy for specificity; subjects with confirmed TB will serve as control group to estimate sensitivity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for PTB, PNTM and extraPTB:

* Adult subjects with documented active pulmonary TB, pulmonary NTM or extrapulmonary TB
* Subjects who have signed informed consent
* Aged ≥18 years

Inclusion criteria for HC:

* healthy donors who have signed informed consent
* aged ≥ 18 years
* no TB or NTM risk factors or exposure

Exclusion Criteria:

Exclusion criteria for PTB, PNTM and extraPTB:

* Do not have active pulmonary TB, NTM or extrapulmonary TB
* Do not sign the informed consent
* Are aged < 18 years

Exclusion criteria for HC:

* Have active pulmonary TB or NTM
* Do not sign the informed consent
* Are aged < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects attending the Infectious Diseases Ward of the participating centers with a pulmonary TB, pulmonary NTM or extrapulmonary TB. Healthy controls,
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic performance of a new test based on the detection of lipoarabinomannan (LAM) antigen in human urine using immunoassay | 12 months
  STANDARDTM F TB LAM Ag FIA is a fluorescent immunoassay for the qualitative detection of specific antigen from mycobacterial lipoarabinomannan (LAM) in urine. The test should be used with the STANDARD F Analyzers manufactured by SD BIOSENSOR that are Europium (Eu) based fluorescent immunoassay system and have been designed for easy and reliable measuring of diverse parameters.
  The test result of a specimen is given either as Positive or Negative with a COI (cut off index) value.
  The test may provide benefits for the development of non sputum-based, less invasive tuberculosis diagnostics that include easier-collect biological samples.
  The results of the test will be compared to the results of the test performed to confirm the pulmonary TB, the extrapulmonary TB or the pulmonary NTM diagnosis Healthy subjects without exposure or risk for TB factors will serve as a proxy for specificity; subjects with confirmed TB will serve as control group to estimate sensitivity.

SECONDARY OUTCOMES:
Exploratory Objectives Evaluate if the test can be used as marker of treatment response (only for PTB subjects) | 6 months
  The test will be repeated at the end of the anti-TB therapy to evaluate if the test can be used as marker of treatment response.We want to evaluate whether, in the face of therapeutic success, the test becomes negative (reversion of results).

CONTACTS AND LOCATIONS:
Locations (1):
- Emerging Bacterial Pathogens Unit, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided